CLINICAL TRIAL: NCT03261323
Title: Evaluating Breast Reconstruction Timing and Risk Reduction Strategies in Patients at a Higher Risk for Developing Breast Reconstruction Surgical Complications: A Prospective Randomized Study
Brief Title: Breast Reconstruction Following Breast Cancer in Very High Risk Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient staff
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE10116
Record Dates: First submitted 2017-07-19; First posted 2017-08-25 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Malignant Neoplasm of Breast
Keywords: Breast Reconstruction; Mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate breast reconstruction (Active Comparator): The surgical schedule will follow unaltered standard protocol for immediate reconstruction right after the patient's mastectomy. Patients will complete a quality of life questionnaire (Breast-Q) both pre-operatively and at different time points during the follow up. The patient's chart will be followed from the mastectomy surgery onwards until 1 year post-final reconstructive surgery for determining complications and hospital costs.
  Interventions: Procedure: Immediate Breast Reconstruction; Other: Breast-Q questionnaire
- Delayed breast reconstruction (Experimental): Patients will start the reconstruction process after cancer therapy has been completed. Patients will be directed to smoking cessation and weight loss resources such as the Bariatric Institute to most directly facilitate risk reduction goals. Risk scores will be assessed at a plastic surgery appointment every 3 months. Reconstruction will proceed after the cancer treatment has been completed, according to individual patient evaluation. Patients will complete a quality of life questionnaire (Breast-Q) both pre-operatively and after the final reconstruction surgery. The patient's chart will be followed from the mastectomy surgery onwards until 1 year post-final reconstructive surgery for determining complications and hospital costs.
  Interventions: Procedure: Delayed Breast Reconstruction; Other: Breast-Q questionnaire

INTERVENTIONS:
Procedure: Immediate Breast Reconstruction — Only implant based surgeries will be considered in this study. The patient will be followed for at least 1 year after the last reconstruction surgery. Reconstruction will be attempted immediately after mastectomy.
  Arms: Immediate breast reconstruction
Procedure: Delayed Breast Reconstruction — Risk reduction strategies on smoking, weight, and chronic disease control will be offered. The individual risk will be recalculated every three months. Delayed breast reconstruction will be offered when core cancer therapies (mastectomy, chemotherapy and radiation) are complete. Only implant based surgeries will be considered in this study. The patient will be followed for at least 1 year after the last reconstruction surgery.
  Arms: Delayed breast reconstruction
Other: Breast-Q questionnaire — Developed out of Memorial Sloan-Kettering Institute for Cancer Research, this questionnaire is designed to create a patient-reported outcome measure to provide quantifiable information about the impact and effectiveness of breast surgery. In this study it will be used for quality of life assessment

SUMMARY:
The purpose of this study is to:

1. Evaluate whether immediate or delayed reconstruction should be offered for breast reconstruction candidates with higher risk for surgical complications by comparing complications, quality of life, and hospital costs
2. Determine the efficacy of risk reduction strategies for breast reconstruction patients with higher risk for surgical complications

DETAILED DESCRIPTION:
Primary Endpoint(s)

1. Define the optimal timing of reconstruction in patients at a higher risk for developing breast reconstruction surgical complications through a randomized prospective cohort
2. Compare immediate and delayed reconstruction outcome metrics through retrospective review

Secondary Endpoint(s)

1. Evaluate Quality of life of patients at a higher risk for developing breast reconstruction surgical complications undergoing immediate versus delayed reconstruction.
2. Compare complications and reoperations between immediate versus delayed reconstruction.
3. Compare the hospital costs between immediate versus delayed reconstruction
4. Evaluate the effectiveness of risk reduction strategies

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed breast cancer or indication for prophylactic mastectomy.
* Subjects must be breast reconstruction candidates using implant based breast reconstruction.
* Subjects must have a pre-operative risk >20% complication prediction from the Breast Reconstruction Risk Assessment (BRA) Score for implant-based breast reconstruction candidates
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior breast cancer surgical treatment
* Prior breast reconstruction
* Inability to provide written consent

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
optimal timing of reconstruction in patients at a higher risk for developing breast reconstruction surgical complications | Until 1 year post breast reconstruction
  Proportion of patients preferring delayed reconstruction.

SECONDARY OUTCOMES:
Major complications | Until 1 year post breast reconstruction
  defined as the ones that required reoperation (infection, capsular contracture, hematoma, seroma, skin flap and flap necrosis, etc).
Minor complications | Until 1 year post breast reconstruction
  defined as the ones that were office treated, not requiring a reoperation
Number of revision surgeries | Until 1 year post breast reconstruction
  defined as surgeries not related to complications, indicated for symmetrization, aesthetic improvement, nipple reconstruction, or skin paddle removal
Hospital cost of the complete reconstruction treatment | Until 1 year post breast reconstruction
  Cost of reconstruction including the cost of complications
Change in patient satisfaction | Until 1 year post breast reconstruction
  Patient satisfaction using the pre-operative Breast-Q questionnaire to define the baseline compared to score on Breast-Q questionnaire during follow-up

OTHER OUTCOMES:
Aesthetic evaluation | Until 1 year post breast reconstruction
  Aesthetic evaluation using postoperative photos one year after the first surgery, and after the final reconstruction surgery

CONTACTS AND LOCATIONS:
Overall Officials: Risal Djohan, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States